CLINICAL TRIAL: NCT01088529
Title: A Randomized, Open-Label, Neoadjuvant Prostate Cancer Trial of Abiraterone Acetate Plus LHRHa Versus LHRHa Alone
Brief Title: Neo-adjuvant Abiraterone + Luteinizing Hormone-Releasing Hormone (LHRH) Versus LHRH in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016945; COU-AA-203 (Other: Cougar Biotechnology, Inc.)
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Cancer
Keywords: Neoadjuvant Prostate Cancer; Abiraterone Acetate; LHRHa; high risk prostate cancer; Radical prostatectomy; Prednisone; Luteinizing Hormone-Releasing Hormone; LHRH analogue
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AA+LHRHa (Experimental): Participants received luteinizing hormone-releasing hormone analog (LHRHa) for a maximum of 4 months (monthly injection or injection every 3 months) and 1,000 mg abiraterone acetate (AA) plus 5 mg of prednisone daily for 3 months prior to radical prostatectomy.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone; Drug: LHRHa
- LHRHa (Experimental): Participants received luteinizing hormone-releasing hormone analog (LHRHa) for a maximum of 4 months (monthly injection or injection every 3 months) prior to radical prostatectomy.
  Interventions: Drug: LHRHa

INTERVENTIONS:
Drug: Abiraterone Acetate — 1000 mg oral daily for 3 months followed by a prostatectomy.
  Other Names: CB7630
  Arms: AA+LHRHa
Drug: Prednisone — 5 mg orally daily.
  Arms: AA+LHRHa
Drug: LHRHa — LHRH analogue (either leuprolide or goserelin): Leuprolide is an intramuscular injection, and goserelin subcutaneous (under skin) of abdomen, given either 1 injection every 3 months or 1 injection each month for 3 months.
  Other Names: Lupron®; leuprolide; Zoladex®; goserelin

SUMMARY:
The goal of this clinical research study is to find out how treatment with abiraterone acetate in combination with prednisone and a Luteinizing Hormone-Releasing Hormone (LHRH) analogue changes the tumor in comparison to treatment with an LHRH analogue alone.

Objectives:

Primary Objective:

To assess the difference in pathologic stage < pT2 between Group A and Group B.

Secondary Objective:

* To assess and compare the changes in levels of androgens (pre, during, and post treatment) in the serum, primary tumor microenvironment and bone marrow between Group A and Group B.
* To assess changes in biomarkers related to androgen signaling and other cancer-related pathways between Group A and Group B.
* To assess the difference in rate of positive surgical margins between Group A and Group B.
* To assess the safety profile of abiraterone acetate and low dose prednisone in a preoperative setting.

DETAILED DESCRIPTION:
Study Groups:

Participants who are eligible to take part in this study will be randomly assigned (as in the flip of a coin) to 1 of 2 groups:

* Those who are in Group A will take abiraterone acetate, a LHRH analogue, and prednisone.
* Those who are in Group B will receive a LHRH analogue alone. Participants will have 2 out of 3 chances of being placed in Group A or 1 out of 3 chances of being placed in Group B.

Participants in both groups will receive the study drug(s) for about 3 months followed by a prostatectomy (prostate surgery) between 2 and 4 weeks after they stop taking the study drug(s).

Length of Study:

Participants will receive study drugs on this study for about 3 months before having surgery to remove their prostate about 2-4 weeks later. Participants will be removed from this study if the disease gets worse, if they experience intolerable side effects, or their study doctors feel that it is in their best interest to stop the study.

Long-Term Follow-Up:

Participants will return to the clinic 1 month, 3 months, 6 months, and then every 6 months (for up to 8 years) after your surgery for follow-up visits. Up to 66 patients will be take part in this study. All will be enrolled at M. D. Anderson after their surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proof of prostatic adenocarcinoma via a minimum of 6 core biopsy samples
2. Clinical stage T1c or T2 with high-grade disease (Gleason's 8-10) on initial biopsy, or clinical stage T2b-T2c with Gleason's grade >/= 7 and PSA > 10ng/ml.
3. No evidence of metastatic disease as determined by CT scans and bone scans.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of </= 1
5. Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (ANC) > 1,500 and platelet count of > 100,000.
6. Normal pituitary and adrenal function
7. Patients should be deemed to be candidates for radical prostatectomy.

Exclusion Criteria:

1. Histological variants in the primary tumor (histological variants other than adenocarcinoma); neuroendocrine tumor
2. Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
3. Uncontrolled hypertension
4. Abnormal Liver function
5. Active or symptomatic viral hepatitis or chronic liver disease
6. Clinically significant heart disease
7. Other active malignancy
8. History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
9. Previous treatment with abiraterone acetate
10. Patients who are not appropriate surgical candidates for radical prostatectomy
11. Prior chemotherapy or radiation therapy for prostate cancer.
12. Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study

Note: There are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc. Clinical Trial, Study Director — Cougar Biotechnology, Inc.; Christopher Logothetis, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- Houston, Texas, United States

REFERENCES:
- See also: NATIONAL CANCER INSTITUTE — http://www.cancer.gov
- See also: NATIONAL INSTITUTE OF HEALTH — http://www.nlm.nih.gov/medlineplus/prostatecancer.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 20 November 2009 to 14 March 2013. Participants were recruited at 1 study center in the United States.
Pre-assignment Details: 66 participants were randomly allocated to the 2 treatment arms and were included in the intent-to-treat (ITT) analysis set. 65 participants received at least 1 dose of the study drug and were included in the safety analysis set.
Period: Overall Study
Arm/Group | AA+LHRHa | LHRHa
Started | 44 | 22
Received Treatment | 44 | 21
Completed | 44 | 21
Not Completed | 0 | 1
Not completed — Did not receive study treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AA+LHRHa | LHRHa | Total
Number analyzed (Participants) | 44 | 22 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (7.14) | 59.9 (7.6) | 61 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 44 | 22 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Pathology Tumor Stage of Less Than or Equal to Prostate Cancer Stage at Which the Tumor is Confined to the Prostate (pT2)
Description: The table below shows number of participants in each treatment group with a pathology tumor stage less than or equal to pT2.
Time Frame: At the end of Cycle 3 (at radical prostatectomy)
Population: Intent-to-treat (ITT) analysis set, which included all participants who were randomized to study.
Measure: Number; unit: participants
Arm/Group | AA+LHRHa | LHRHa
Number analyzed (Participants) | 44 | 22
participants | 24 | 8
Statistical Analysis 1: Comparison: AA+LHRHa vs LHRHa; Test type: Superiority or Other; p = 0.2148, Chi-squared; Relative risk = 1.432, 90% CI 2-sided [0.859 to 2.386]

2. Secondary Outcome: Number of Participants With a Positive Surgical Margin at Radical Prostatectomy
Description: The table below shows number of participants in each treatment group who had positive surgical margins. A positive surgical margin is defined as tumor extending to the inked-surface or margin of the prostate.
Time Frame: At the end of Cycle 3 (at radical prostatectomy)
Population: Intent-to-treat (ITT) analysis set, which included all participants who were randomized to study.
Measure: Number; unit: participants
Arm/Group | AA+LHRHa | LHRHa
Number analyzed (Participants) | 44 | 22
participants | 6 | 6
Statistical Analysis 1: Comparison: AA+LHRHa vs LHRHa; Test type: Superiority or Other; p = 0.1796, Fisher Exact; Relative risk = 0.477, 90% CI 2-sided [0.205 to 1.109]

3. Secondary Outcome: Number of Participants With Prostate-Specific Antigen Response
Description: The table below shows number of participants in each treatment group who achieved a prostate-specific antigen (PSA) response defined as a drop in PSA value to less than or equal to 0.2 ng/mL.
Time Frame: Cycle 3 Day 1
Population: Intent-to-treat (ITT) analysis set, which included all participants who were randomized to study. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | AA+LHRHa | LHRHa
Number analyzed (Participants) | 44 | 20
participants | 32 | 0
Statistical Analysis 1: Comparison: AA+LHRHa vs LHRHa; Test type: Superiority or Other; p < 0.0001, Chi-squared; Relative risk = 6.523, 90% CI 2-sided [2.701 to 15.753]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | AA+LHRHa | LHRHa
Serious Adverse Events (participants affected / at risk) | 2/44 | 2/21
Other Adverse Events (participants affected / at risk) | 43/44 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AA+LHRHa (N=44) | LHRHa (N=21)
Gastric Ileus (Gastrointestinal disorders) | 0 | 1
Infected Lymphocele (Infections and infestations) | 1 | 0
Pelvic Abscess (Infections and infestations) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AA+LHRHa (N=44) | LHRHa (N=21)
Anaemia (Blood and lymphatic system disorders) | 23 | 8
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 4 | 2
Fatigue (General disorders) | 19 | 10
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 1
Alanine Aminotransferase Increased (Investigations) | 22 | 7
Aspartate Aminotransferase Increased (Investigations) | 17 | 7
Blood Sodium Increased (Investigations) | 1 | 2
Blood Urea Increased (Investigations) | 0 | 2
Blood Uric Acid Increased (Investigations) | 3 | 1
Platelet Count Decreased (Investigations) | 4 | 0
White Blood Cell Count Decreased (Investigations) | 3 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Cognitive Disorder (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 6
Pollakiuria (Renal and urinary disorders) | 3 | 0
Urinary Incontinence (Renal and urinary disorders) | 3 | 3
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 2
Hot Flush (Vascular disorders) | 37 | 18
Hypertension (Vascular disorders) | 10 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days